CLINICAL TRIAL: NCT07262216
Title: Correlation Between Pain Threshold and Analgesic Consumption During Egg Collection in Patients
Brief Title: Correlation Between Pain Threshold and Analgesic Consumption in Transvaginal Oocyte Aspiration Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Burcu ayvazoğlu (Other)
Responsible Party: Sponsor-Investigator, Burcu ayvazoğlu, research assistant, TC Erciyes University
Organization: TC Erciyes University (Other)
Other Study IDs: Erciyes university medical sch
Record Dates: First submitted 2025-05-15; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Pain Threshold; Conscious Sedation; Oocyte Retrieval
Keywords: Oocyte retrieval; conscious sedation; Pain threshold

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Nowadays, in vitro fertilization (IVF) is an important component of modern infertility treatment. One of the critical stages of the IVF process is oocyte (egg) retrieval, which requires both anesthesia and analgesia; this directly affects the comfort of the participants and the success of the procedure. Since its first implementation, various methods and techniques have been used for oocyte retrieval, and today it is most commonly performed under anesthesia with transvaginal ultrasonography guidance.

Because this procedure is performed on an outpatient basis in IVF centers worldwide, the anesthetic agents used are expected to meet several essential criteria: they should have a short half-life, a rapid onset of action, and minimal, acceptable side effects. In addition, these agents should not adversely affect participants' recovery processes. While the agents used determine the quality of sedation and analgesia, concerns persist regarding their potential negative effects on reproductive outcomes.

Considering that participants often experience high levels of anxiety, effective pain management must be ensured during the procedure. Moreover, participants must remain immobile throughout the procedure. To achieve this, general anesthesia, regional/local anesthesia, neuraxial anesthesia, patient-controlled analgesia, sedation, acupuncture, or combinations of these methods may be used.

Conscious sedation is the most commonly applied anesthesia method for women undergoing transvaginal oocyte aspiration. This method is preferred by approximately 95% of IVF centers in the USA and 84% in the UK. Conscious sedation allows the participant to maintain airway control and adequate oxygenation independently, while also providing a reduction in consciousness.

Currently, midazolam, propofol, and fentanyl are the most frequently preferred agents for this purpose. They are easy to administer and are safe for cooperative participants. Compared to other anesthetic agents, they have relatively lower negative effects on oocyte and embryo quality and fewer adverse impacts on pregnancy rates. However, studies have shown that midazolam, fentanyl, and alfentanil can be detected in follicular fluid even after a single dose. In vitro studies on mouse oocytes and some human studies have indicated that propofol may have dose-dependent harmful effects on fertilization. Therefore, some researchers recommend that propofol should be used with caution during oocyte retrieval, with attention to limiting the total dose administered. As prolonged exposure to anesthetic agents has been shown to negatively affect fertilization, it is recommended that oocytes be exposed to anesthetic agents at the lowest possible level. Thus, for successful outcomes, it is critical that the anesthetic agents used during transvaginal follicle aspiration be administered at appropriate doses and durations.

The researchers aim in this study to examine the correlation between the amount of anesthetic agent required and the pain threshold in participants whose pain thresholds are measured and who receive patient-controlled analgesia combined with conscious sedation. As a secondary objective, the researchers aim to compare participants' demographic characteristics, sociocultural status, stress and anxiety levels, the amount of anesthetic agent used, and its hemodynamic effects.

This study is designed as a prospective, open-label, single-arm, non-randomized study. Forty female participants aged 18-50 years who will undergo oocyte retrieval for IVF treatment at the Erciyes University Department of Obstetrics and Gynecology will be included. To assess participants' pre-procedural stress and anxiety levels, the Spielberger State-Trait Anxiety Inventory (STAI) will be administered. Each participant's pain threshold will be measured at three sites-one muscle area (deltoid) and two bony areas (thumb and mid-tibia)-using an algometer (Commander Echo Algometer, JTECH Medical, Midvale, UT, USA), with bilateral measurements taken once at each site. The average of these three measurements will be calculated to determine the overall body pressure pain threshold for each participant.

Prior to the procedure, all participants will receive 1.5 mg midazolam IV. During conscious sedation, a pre-prepared solution of 15 cc 1% propofol (150 mg) and 5 cc fentanyl (250 mcg) in a total volume of 20 cc will be administered using a PCA device with no lockout interval. Participants will be instructed to press the PCA button whenever they begin to feel pain. Hemodynamic parameters (systolic, diastolic, and mean arterial pressure, heart rate, SpO₂), Ramsay Sedation Scale (RSS) and Facial Score (FS) values will be recorded throughout the procedure. After the procedure, participants will be closely monitored for nausea, vomiting, and respiratory depression. In addition, total follicle count, embryo count, and pregnancy status will be recorded

DETAILED DESCRIPTION:
e English academic translation of your text:

In vitro fertilization (IVF) is a promising treatment modality that provides infertile couples with the opportunity to conceive, and its success rates have continued to increase with technological advancements. The IVF treatment process consists of four fundamental stages: ovarian stimulation, oocyte retrieval, fertilization, and embryo transfer. Ultrasound-guided transvaginal oocyte aspiration is considered the gold standard for oocyte retrieval.

Pain is commonly experienced during transvaginal oocyte aspiration, necessitating the use of anesthesia. IVF procedures are typically performed in outpatient settings within assisted reproduction centers. The ideal anesthetic technique in IVF should have minimal side effects, ensure a rapid recovery, provide high pregnancy rates, and offer both patient and surgical team comfort and safety. Many anesthetic agents used during IVF have been detected in follicular fluid. These agents may potentially influence fertilization, implantation, and embryo quality, thereby affecting treatment success. However, studies investigating the effects of anesthetics on fertilization and embryo quality have yielded inconsistent and inconclusive results.

A variety of anesthesia techniques can be employed during transvaginal oocyte aspiration, including general anesthesia, regional/local anesthesia, neuraxial anesthesia, patient-controlled analgesia, sedation, acupuncture, or combinations of these modalities.

A study published in 2023 that reviewed literature from 1987 to 2022 reported that conscious sedation was the most frequently preferred anesthetic technique for women undergoing transvaginal oocyte aspiration. This approach was associated with fewer side effects, faster recovery, higher patient and physician satisfaction, and fewer adverse effects on oocyte and embryo quality. High levels of patient satisfaction have been reported with this method.

During oocyte retrieval, patients experience pain due to needle puncture of the vaginal wall and ovaries and due to manipulation of the aspiration needle. Various opinions exist regarding the nature of this pain. In a study by Wicke et al. involving 277 patients, analgesic administration significantly reduced pain severity during the procedure (mean pain score was 1.21 in patients receiving analgesia vs. 9.26 in those who did not). Younger patients and those with a history of dysmenorrhea reported higher pain scores compared to others.

The IVF treatment process is also associated with considerable psychological stress. Most patients undergoing IVF are over the age of 30 and may have chronic medical conditions, experience familial pressure, and be predisposed to depression or psychosis. Hormonal treatments administered during the process can further exacerbate these symptoms. These medical and psychological factors collectively increase patient anxiety. Therefore, anesthesiologists must be capable of managing preoperative anxiety, which can be assessed using validated questionnaires.

With the approval of Erciyes University Faculty of Medicine Clinical Research Ethics Committee (approval number: 2024/275), the study entitled "Correlation between Pain Threshold and Analgesic Consumption during Oocyte Retrieval: An Open-label, Single-arm, Non-randomized Study" will be conducted at Erciyes University Department of Obstetrics and Gynecology. Exclusion criteria include a history of dyspareunia, major medical or psychiatric disorders, and vaginismus.

Before the procedure, patients will be informed by an anesthesiologist about the process, conscious sedation, and the patient-controlled analgesia (PCA) device. The State-Trait Anxiety Inventory (STAI) will be administered to evaluate pre-procedural stress and anxiety levels. Patients will complete the questionnaire either independently or with assistance from the anesthesiologist. Written informed consent will be obtained.

Pain threshold will be measured using a digital algometer routinely used in clinical settings (Commander Echo Algometer, JTECH Medical, Midvale, UT, USA), which allows measurements in kilograms, pounds, or Newtons. The device has been validated in previous studies. The examiner will hold the algometer with the right hand while supporting the device with the left hand. To familiarize patients with the sensation of pressure, an initial application will be performed on a non-test area (thenar region). Patients will be instructed to say "stop" when the pressure sensation turns into pain. Pressure will be applied at a constant rate of 1 kg/s and a 90° angle until the patient gives the stop command. This familiarization will be performed three times per patient. All measurements will be conducted by the same operator, in the same room, at a consistent ambient temperature, using the same equipment. A 1 cm² probe will be used, and measurements will be recorded in kg/cm². Each anatomical region will be measured bilaterally in a fixed order, with three measurements taken at 5-second intervals. The average of the three values will be recorded as the pain threshold for each site. Measurements will be taken from one muscular site (deltoid) and two bony sites (thumb and mid-tibia). For deltoid measurements, the patient will be seated with the arm resting beside the torso and the elbow in extension; measurements will be taken 2 cm distal to the acromion. For thumb measurements, the thumb will rest volar side down on a table, excluding MCP and IP joints, with the wrist in neutral position. For tibia measurements, patients will sit with feet flat and knees flexed to 60°, and pressure will be applied 6 cm distal to the tibial tuberosity. The average of the three values from each site will be calculated, and a global pressure pain threshold will be derived.

In the operating room, routine monitoring will include electrocardiography (ECG), peripheral oxygen saturation (SpO₂), and noninvasive blood pressure. Patients will be placed in the lithotomy position, and oxygen will be delivered via nasal cannula at 2-4 L/min. Demographic data (height, weight, education level), ASA classification, procedure duration, and intraoperative hemodynamic parameters will be recorded. Hemodynamic parameters including systolic, diastolic, and mean arterial pressures (SAP, DAP, MAP), heart rate (HR), and SpO₂ will be recorded at baseline and at 5, 10, 15, and 20 minutes.

Facial Scale (FS) scores ranging from 0 (no pain) to 5 (very severe pain) will be used by the anesthesiologist to assess facial expressions at 5, 10, 15, and 20 minutes. Ramsay Sedation Scale (RSS) scores will be recorded at the same intervals, ranging from 1 (anxious, agitated) to 6 (no response to painful stimuli).

Five minutes prior to the procedure, 1.5 mg IV midazolam (Sedever®) will be administered. Conscious sedation will be provided via PCA, prepared using 150 mg (15 ml) propofol 1% (Propofol-PF®) and 250 µg (5 ml) fentanyl (Fentanyl-PF®), diluted to 20 ml. Each bolus will contain 2 ml (15 mg propofol + 25 µg fentanyl), without a lock-out interval. Patients will be instructed to press the PCA button upon feeling pain, allowing self-titration of anesthesia to avoid excessive anesthetic exposure and potential harm to oocyte quality.

Desaturation is defined as SpO₂ <92% for more than 10 seconds. Bradycardia is defined as HR <50 bpm; tachycardia as a >20% increase from baseline. Hypotension and hypertension are defined as MAP values 20% below or above baseline, respectively.

Postoperatively, patients will be monitored in the recovery unit for nausea, vomiting, and respiratory depression. Complications will be recorded. Once discharge criteria are met, both patient and surgeon satisfaction will be assessed. Pregnancy status, total number of follicles, and number of embryos will also be recorded post-procedure

ELIGIBILITY:
Inclusion Criteria:

* Women receiving IVF treatment

Exclusion Criteria:

* Dyspareunia history
* Psychiatric disease
* Vaginismus
* ASA 3 patients

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Study Population: Women who applied to the IVF center for treatment and agreed to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-12-08 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the correlation between the pre-procedural pain threshold measured in kg/cm² with an algometer and the amount of anesthetic agents used during the procedure in IVF patients undergoing conscious sedation | 1 day
  In this study, the researchers aimed to examine the relationship between the pre-procedurally measured pain threshold and the amount of anesthetic agent required during patient-controlled analgesia and conscious sedation; in this specific group of patients undergoing IVF treatment, where potential adverse effects of anesthetic agents on oocytes are avoided, we aimed to evaluate the correlation between pain threshold values measured in kg/cm² using an algometer and the amount of anesthetic agents administered during the procedure.

SECONDARY OUTCOMES:
Age | 1 day (will be recorded before the process begins)
  This result will evaluate the relationship between the age of the participants (years) and the amount of anesthetic used during the procedure.
Body Mass Index | 1 day (will be recorded before the process begins)
  This output will assess the relationship between participants' body mass index (kg/m²) and the amount of anesthetic used during the procedure
Spielberger State-Trait Anxiety Inventory Score | 1 day (will be recorded before the process begins)
  This output will assess the relationship between participants' Spielberger State-Trait Anxiety Inventory scores and the amount of anesthetic used during the procedure.
Educational Status | 1 day (will be recorded before the process begins)
  This output will assess anesthetic use by participants at different educational levels (primary school, secondary school, university)

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes üniversitesi tıp fakültesi hastanesi, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes